CLINICAL TRIAL: NCT04217980
Title: Analysis of a Diagnostic Algorithm of Severe Pneumonia in Pediatric Critical Patients by Pulmonary Ultrasound and Procalcitonin as a Plan to Improve the Quality of Care
Brief Title: Severe Pneumonia Diagnostic in Pediatric Population by Lung Ultrasonography and Procalcitonin
Acronym: PROLUSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: FSJD-NEUMO-2017
Record Dates: First submitted 2019-12-03; First posted 2020-01-06 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Pneumonia Childhood
Keywords: pneumonia; lung ultrasound; biomarkers; procalcitonin; childhood
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung ultrasonography (LUS) group (Experimental): Group 1: Lung ultrasonography is performed as the main (first) pulmonary image test
  Interventions: Diagnostic Test: Lung ultrasonography (LUS) or Chest X ray (CXR)
- Chest X ray (CXR) group (Active Comparator): Group 2: Chest X ray is performed as main (first) pulmonary image test
  Interventions: Diagnostic Test: Lung ultrasonography (LUS) or Chest X ray (CXR)

INTERVENTIONS:
Diagnostic Test: Lung ultrasonography (LUS) or Chest X ray (CXR) — pediatrician researcher (PR) will conduct a LUS or CXR at admission time as a first test of lung image depending on randomized group.

SUMMARY:
Lung ultrasound (LUS) in combination with a biomarker has not yet been studied. The investigators propose a clinical trial where the primary aims are: 1. To assess whether an algorithm with LUS and procalcitonin (PCT) may be useful for diagnosing bacterial pneumonia; 2. To analyse the sensitivity and specificity of LUS vs chest radiograph (CXR).

DETAILED DESCRIPTION:
Objectives: The general objective is to analyze whether a new algorithm approach of severe pneumonia in pediatric intensive unit (PICU) improves the quality of care. Objectives: 1- To analyze the sensitivity and specificity of lung ultrasound (LUS) compared respect to the chest radiography (CXR) in severe pneumonia and if LUS discriminates between bacterial and viral one. 2- If there is a lower CXR indication. 3- If is possible to reduce the dose of irradiation and costs associated with CXR. 4- To analyze the interobserver agreement of the LUS. 5- determine whether a diagnosis of pneumonia algorithm using LUS and procalcitonin may be useful in directing the indication of antibiotic therapy and / or the duration thereof.

Methodology: clinical, prospective, controlled, randomized, blinded intervention and 3-year trial. Inclusion of children under 18 years, with severe pneumonia, who enter (PICU). Experimental Group 1: pediatrician researcher (PR) will conduct a LUS at admission time, as a first test of lung image; in Group 2, CXR is conduced as first image. Patients will be classified into 3 subgroups, in both branches: a) if PCT is <1 ng /L and LUS is not suggestive of bacterial pneumonia, no antibiotic will be prescribed; b) if LUS is suggestive of bacterial pneumonia, regardless of the PCT, it will be recommended to start antibiotic therapy; c) If the ultrasound is suggestive of bacterial pneumonia but PCT is> 1 ng / L, antibiotic therapy will be recommended to cover other causes of infection. The same attitude will be performed, but depending on the CXR instead of the LUS, in group 2. Clinical variables, complementary tests and evolution data will be collected. Statistics by SPPS® 20.0. Informed consent will be requested and the study will be conducted according to the Helsinki Declaration guidelines and Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* children under 18
* severe pneumonia criteria
* admitted at PICU
* informed consent signed

Exclusion Criteria:

* previous respiratory disease (cystic fibrosis and/or immunosuppression)
* Nosocomial pneumonia development while in charge for community pneumonia.
* Researcher pediatrician has valuated the chest X ray before the PICU admission
* Included in other clinical trial

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 202 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Sensibility and specificity of LUS and procalcitonin for pneumonia diagnosis | through study completion, an average of 2 years
  Sens and Spe for LUS group and for X-Ray group

SECONDARY OUTCOMES:
antibiotic days of treatment | through study completion, an average of 2 years
  antibiotic duration for CXR group and antibiotic duration for LUS group

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Fundació Sant Joan de Déu, Esplugues de Llobregat

REFERENCES:
- [Derived] Guitart C, Bobillo-Perez S, Rodriguez-Fanjul J, Carrasco JL, Brotons P, Lopez-Ramos MG, Cambra FJ, Balaguer M, Jordan I. Lung ultrasound and procalcitonin, improving antibiotic management and avoiding radiation exposure in pediatric critical patients with bacterial pneumonia: a randomized clinical trial. Eur J Med Res. 2024 Apr 6;29(1):222. doi: 10.1186/s40001-024-01712-y. PMID 38581075
- [Derived] Rodriguez-Fanjul J, Guitart C, Bobillo-Perez S, Balaguer M, Jordan I. Procalcitonin and lung ultrasound algorithm to diagnose severe pneumonia in critical paediatric patients (PROLUSP study). A randomised clinical trial. Respir Res. 2020 Oct 8;21(1):255. doi: 10.1186/s12931-020-01476-z. PMID 33032612